CLINICAL TRIAL: NCT06082856
Title: Evaluation of the Hemodynamic Effect of Dexmedetomidine in Scheduled Outpatient Surgery: Single-center Prospective Randomized Double-blind Non-inferiority Study.
Brief Title: Evaluation of the Hemodynamic Effect of Dexmedetomidine in Scheduled Outpatient Surgery
Acronym: DEXCOEUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NIMAO/2022-1/YG01
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Dexmedetomidine; Hemodynamics; Ambulatory Care
MeSH Terms: interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Sufentanil (Active Comparator)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Induction of general anesthesia by administration of dexmedetomidine 0.5µg/Kg (maximum dose 50 µg) in titration by bolus of 10µg intravenously over 5 minutes
  Arms: Dexmedetomidine
Drug: Sufentanil — Induction of general anesthesia by administration of sufentanil 0.25µg/Kg (maximum dose 20 µg) intravenously at anesthetic induction.
  Arms: Sufentanil

SUMMARY:
Ambulatory surgery is increasingly used in anesthesia. In case of general anesthesia, it is recommended to use anesthesia molecules with a short half-life and low doses of opiates to ensure a rapid awakening and to prevent nausea and vomiting by systematic administration of anti-emetics during the operation.

Opiates (including sufentanil) have recently been called into question because of the nausea and vomiting and the delay in waking up induced by these molecules. To combat these side effects, the authors have proposed either to reduce the doses or to substitute them with dexmedetomidine, a sedative antihypertensive drug. Recent studies have demonstrated that opiates used in general anesthesia can be replaced by dexmedetomidine. However, literature data are controversial concerning the hemodynamic impact. No study has compared the hemodynamic profile of opioid-free anesthesia with dexmedetomidine versus conventional anesthesia with opioids.

The ambulatory context lends itself to the use of dexmedetomidine because it is aimed at a population without strong cardiac pathology, concerns non-major interventions, with the need to optimize pain and side effects.

The study authors therefore wish to compare the effects of induction of general anesthesia with low-dose Dexmedetomidine versus sufentanil, on post-induction hemodynamic stability in scheduled outpatient surgeries. The investigators hypothesize that hemodynamic stability at induction of general anesthesia with low-dose dexmedetomidine is not inferior to that obtained with sufentanil in scheduled ambulatory surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patient with scheduled surgery under general anesthesia for one of the following: oral, orthopedic, urological, digestive and gynecological surgeries.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study
* The subject is unable to give consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient with a known allergy to dexmedetomidine or other drugs.
* Patient with a contraindication to general anesthesia or outpatient management.
* Patient treated with beta-blocker, ACE inhibitor or ARB2
* Patient with an ASA4 score.
* Patient with HR < 50 bpm.
* Patient with the following cardiovascular comorbidities: coronary insufficiency, obstructive cardiomyopathy, severe hypertension, ventricular rhythm or conduction disorder.
* Patient with hepatic (prothrombin rate < 70%, liver enzyme/Bilirubin X 3) and/or renal (clearance < 50 ml.min) insufficiency.
* Pregnant, parturient or nursing patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hemodynamic stability during anesthesia between groups | Within 60 minutes after induction
  Incidence of mean arterial pressure < 60 mmHg

SECONDARY OUTCOMES:
Intraoperative hemodynamic stability according to baseline mean arterial pressure between groups | Within 60 minutes after induction
  Percentage of patients with 30% change in mean arterial pressure from baseline
Intraoperative heart rate between groups | Within 60 minutes after induction
  Percentage of patients with bradycardia ≤45bpm/min
Intraoperative hypertensive episodes between groups | Within 60 minutes after induction
  Percentage of patients with at least one episode of arterial hypertension (mean arterial pressure > 100mmHg)
Hemodynamic stability in the ICU between groups | Day 0 at discharge from ICU
  Percentage of patients with at least one episode of a Systolic Blood Pressure below 90mmHg (SBP < 90mmHg) in the ICU
Intraoperative vasopressor use between groups | Day 0, during surgery
  Amount of IV Ephedrine (in mg) administered intraoperatively to maintain mean arterial pressure > 60 mmHg
Intraoperative IV Atropine use between groups | Day 0, during surgery
  Amount of IV Atropine (in µg) administered intraoperatively to maintain a heart rage > 45bpm
Failure of ambulatory management between groups between groups | Day 1
  Percentage of patients hospitalized after surgery
Patient reported pain between groups | Day 0
  Pain reported on a 0-10 visual analog scale
Patient reported pain between groups | Day 1
  Pain reported on a 0-10 visual analog scale
Patient reported pain between groups | Day 2
  Pain reported on a 0-10 visual analog scale
Patient reported pain between groups | Day 7
  Pain reported on a 0-10 visual analog scale
Immediate nausea and vomiting between groups | Day 0 during ICU stay
  Percentage of patients with nausea and vomiting according to use of Ondansetron IV
Post-operative nausea and vomiting between groups | Day 0 at discharge from surgery
  Percentage of patients reporting absence/presence nausea and vomiting
Post-operative nausea and vomiting between groups | Day 1
  Percentage of patients reporting absence/presence nausea and vomiting
Post-operative nausea and vomiting between groups | Day 2
  Percentage of patients reporting absence/presence nausea and vomiting
Post-operative nausea and vomiting between groups | Day 7
  Percentage of patients reporting absence/presence nausea and vomiting
Patient postoperative recovery between groups | Day 2
  Quality of Recovery questionnaire (QoR-40) (score 0-200)
Patient satisfaction with perioperative management between groups | Day 2
  Evaluation of Experience of General Anesthesia questionnaire (EVAN-G) (score 5-100)
Occurrence of adverse events after surgery between groups | Day 2
  Absence/presence of the following adverse events: bleeding, hematoma or re-hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Yann Gricourt, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France